CLINICAL TRIAL: NCT03326973
Title: Long-Term Quality of Life in Patients With Metastatic Melanoma Treated With Checkpoint Inhibitors
Status: Completed | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 17-518
Record Dates: First submitted 2017-10-27; First posted 2017-10-31 (Actual); Last update posted 2020-12-17 (Actual); Status verified 2020-12

CONDITIONS: Metastatic Melanoma
Keywords: Quality of Life (QoL); 17-518
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- online or telephone survey: This is a cross-sectional survey. Our main method of communication with patients will be email. Participants will complete a single online or telephone survey at a minimum of 12 months post initial treatment of checkpoint inhibitors and remain on maintenance therapy.
  Interventions: Behavioral: EuroQoL EQ-5D-3L; Behavioral: EORTC QLQ-C30; Other: PRO-CTCAE; Behavioral: Fatigue severity score questionnaire; Behavioral: The COST; Behavioral: Physician information

INTERVENTIONS:
Behavioral: EuroQoL EQ-5D-3L — Overall QOL
Behavioral: EORTC QLQ-C30 — General symptoms; physical, role, emotional, cognitive, and social functioning scales; fatigue, nausea/vomiting , and pain scales
Other: PRO-CTCAE — Additional potential immune-specific symptoms
Behavioral: Fatigue severity score questionnaire — Fatigue severity
Behavioral: The COST — Financial toxicity; satisfaction with ability to work
Behavioral: Physician information — Details on outside health providers

SUMMARY:
To identify and describe long-term quality of life (QOL) issues in patients with metastatic melanoma treated with checkpoint inhibitors who achieved cancer control for a minimum of 12 months and remain on maintenance checkpoint inhibitor therapy.

ELIGIBILITY:
Inclusion Criteria:

* Be able to speak and read English
* Be able to provide informed consent
* Have been diagnosed with metastatic melanoma at age 18 years or older
* Have been treated with either single agent or combination checkpoint inhibitor
* Be at least 12 months since first dose of above named agents
* Received no other systemic therapy after initiation of immunotherapy (interval radiation or surgery will be permitted based on review with primary treating medical oncologist)

Exclusion Criteria:

* Patients with cognitive, visual, or motor impairment such that they cannot complete the survey as assessed by the research or clinical team
* Patients who developed a subsequent cancer after starting on checkpoint inhibitor(s), exclusive of non-melanoma superficial skin cancers
* Patients with clinical documentation of progressive disease on the most recent assessment in the electronic medical record
* Patients with symptomatic progression but continue on immunotherapy

  * Note: For any patients where the disease status is not clear, we will confirm that the disease is either stable or responsive with their primary treating medical oncologist

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The melanoma service has agreed to provide this research team with access to a list of patients who are potentially eligible for this survey.
Sampling Method: Non-Probability Sample
Enrollment: 107 (Actual)
Dates: Start 2017-10-25 (Actual); Primary Completion 2020-12-14 (Actual); Study Completion 2020-12-14 (Actual)

PRIMARY OUTCOMES:
total score of Global QOL overall health index | 1 year
  On the EQ-5D-3L, respondents are asked to indicate their health state by marking the box associated with the most appropriate statement in each of the 5 dimensions, resulting in a one digit number expressing the level (1-3) selected for that dimension from no problems to extreme problems.

CONTACTS AND LOCATIONS:
Overall Officials: Deborah Korenstein, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (6):
- United States (6):
  - Memoral Sloan Kettering Basking Ridge, Basking Ridge, New Jersey
  - Memoral Sloan Kettering Monmouth, Middletown, New Jersey
  - Memorial Sloan Kettering Commack, Commack, New York
  - Memorial Sloan Kettering Westchester, Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering Rockville Centre, Rockville Centre, New York

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm